CLINICAL TRIAL: NCT02461524
Title: Endurant Evo International Clinical Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study terminated enrollment due to device failures prior to enrollment completion.
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10173339DOC
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Results first posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2023-09

CONDITIONS: Abdominal Aortic Aneurysm; AAA
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Abdominal Aortic Aneurysm Endovascular repair (Other): Subjects who were appropriate candidates for endovascular repair of infrarenal abdominal aortic or aortoiliac aneurysms and who met the inclusion and exclusion criteria.
  Interventions: Device: Endurant Evo AAA Stent Graft System; Procedure: Endovascular aneurysm repair (EVAR)

INTERVENTIONS:
Device: Endurant Evo AAA Stent Graft System
Procedure: Endovascular aneurysm repair (EVAR)

SUMMARY:
The purpose of this trial is to evaluate the safety and effectiveness of the Endurant Evo Abdominal Aortic Aneurysm (AAA) Stent graft system for endovascular treatment of subjects with infrarenal abdominal aortic or aortoiliac aneurysms.

DETAILED DESCRIPTION:
The Endurant Evo International Clinical Trial is a prospective, multi-center, premarket, non-randomized, single-arm trial.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years old
2. Subject understands and voluntarily has signed and dated the Informed Consent approved by the Sponsor and by the Ethics Committee/Institutional Review Board.
3. Subject is able and willing to comply with the protocol and to adhere to the follow-up requirements
4. Subject is a suitable candidate for elective surgical repair of AAA as evaluated by American Society of Anesthesiologists (ASA) Physical Status Classification System I, II, or III
5. Subject has an infrarenal abdominal aortic or aortoiliac aneurysm characterized by one or more of the following:

   * Aneurysm is > 5 cm in diameter (diameter measured is perpendicular to the line of flow)
   * Aneurysm is 4 - 5 cm in diameter and has increased in size ≥ 0.5 cm within the previous 6 months
6. Subject meets all the following anatomical criteria as demonstrated on contrast-enhanced CT or Magnetic Resonance Angiography (MRA) imaging:

   * Proximal neck length of ≥ 10 mm with ≤ 60° infrarenal and ≤ 45° suprarenal neck angulation or Proximal neck length of ≥ 15 mm with ≤ 75° infrarenal and ≤ 60° suprarenal neck angulation
   * Subject has vascular dimensions, e.g., aortic and iliac diameters, lengths from renal arteries to iliac bifurcation and hypogastric arteries, in the range of sizes available for the Endurant Evo AAA stent graft system (measured intima to intima) and within the sizing recommendations (refer to Endurant Evo AAA stent graft system Instructions for Use (IFU))
   * Subject has a proximal aortic neck diameter ≥18 mm and ≤32 mm
   * The distal fixation center of the iliac arteries must have a diameter ≥7 mm and ≤ 25 mm bilaterally for the bifurcation and unilaterally for the Aorto-Uni-Iliac (AUI)
   * Subject has documented imaging evidence of at least one patent iliac and one femoral artery, or can tolerate a vascular conduit that allows introduction of the Endurant Evo AAA stent graft system
   * Subject has distal non-aneurysmal iliac (cylindrical) fixation length ≥ 20 mm bilaterally for the bifurcation and unilaterally for the AUI

Exclusion Criteria:

1. Subject has a life expectancy ≤ 1 year
2. Subject is participating in another investigational drug or device study which would interfere with the endpoints and follow-ups of this study
3. Subject is pregnant
4. Subject has an aneurysm that is:

   * Suprarenal/ pararenal/ juxtarenal
   * Isolated ilio-femoral
   * Mycotic
   * Inflammatory
   * Pseudoaneurysm
   * Dissecting
   * Ruptured
   * Leaking but not ruptured
5. Subject requires emergent aneurysm treatment
6. Subject has a known, untreated thoracic aneurysm >4.5 cm in diameter at time of screening
7. Subject has been previously treated for an abdominal aortic aneurysm
8. Subject has a history of bleeding diathesis or coagulopathy
9. Subject has had or plans to have an unrelated major surgical or interventional procedure within 1 month before or after implantation of the Endurant Evo AAA stent graft
10. Subject has had a myocardial infarction (MI) or cerebral vascular accident (CVA) within 3 months prior to implantation of the Endurant Evo AAA stent graft
11. Subject has a conical neck defined as a >4 mm distal increase from the lowest renal artery over a 10 mm length
12. Subject has a known allergy or intolerance to the device materials
13. Subject has a known hypersensitivity or contraindication to anticoagulants, antiplatelets, or contrast media, which is not amenable to pre-treatment
14. Subject has significant aortic thrombus and/or calcification at either the proximal or distal attachment centers that would compromise fixation and seal of the device at the discretion of the investigator
15. Subject has ectatic iliac arteries requiring bilateral exclusion of hypogastric blood flow
16. Subject whose arterial access site is not anticipated to accommodate the diameter of the Endurant Evo AAA delivery system (13F-17F) due to vessel size, calcification, or tortuosity
17. Subject is morbidly obese or has other documented clinical conditions that severely inhibit radiographic visualization of the aorta at the discretion of the investigator
18. Subject has active infection at the time of the index procedure documented by e.g. pain, fever, drainage, positive culture and/or leukocytosis considered to be clinically significant per investigator discretion
19. Subject has congenital degenerative collagen disease, e.g., Marfan's Syndrome
20. Subject has a creatinine level >2.00 mg/dl (or >176.8 µmol/L)
21. Subject is on dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2015-06; Primary Completion 2021-06-25 (Actual); Study Completion 2021-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hence Verhagen, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (9):
- Austria (2):
  - Krankenhaus Hietzing, Vienna
  - Wilhelminenspital, Vienna
- Belgium (2):
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven - Campus Gasthuisberg, Leuven
- Odense Universitetshospital, Odense, Denmark
- Netherlands (3):
  - Rijnstate - Locatie Arnhem, Arnhem
  - Catharina Ziekenhuis, Eindhoven
  - Erasmus University Medical Center, Rotterdam
- Skånes Universitetssjukhus Malmö, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened for enrollment based on the study Inclusion/Exclusion criteria between Jun 2015 and Mar 2016.
Groups:
- Endovasculair Repair: Subjects who were appropriate candidates for endovascular repair of infrarenal abdominal aortic or aortoiliac aneurysms and who met the inclusion and exclusion criteria.
Period: Overall Study
Arm/Group | Endovasculair Repair
Started | 69
Completed | 38
Not Completed | 31
Not completed — Death | 16
Not completed — Withdrawal by Subject | 4
Not completed — Device Explanted | 5
Not completed — Missed Visit | 6

BASELINE CHARACTERISTICS:
Groups:
- Abdominal Aortic Aneurysm Endovasculair Repair: Subjects who were appropriate candidates for endovascular repair of infrarenal abdominal aortic or aortoiliac aneurysms and who met the inclusion and exclusion criteria.
Arm/Group | Abdominal Aortic Aneurysm Endovasculair Repair
Number analyzed (Participants) | 69
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.8 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 61
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 34
  Sweden | 9
  Austria | 5
  Belgium | 11
  Denmark | 10

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint Assessed by the Number of Participants Experiencing a Major Adverse Event (MAE) Within 30-days Post-implantation.
Description: MAEs include the occurrence of any of the following events:
  All-cause mortality Bowel ischemia Myocardial infarction Paraplegia Procedural blood loss ≥1000 cc Renal failure Respiratory failure Stroke
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal Aortic Aneurysm Endovascular Repair
Number analyzed (Participants) | 69
Participants | 2
Statistical Analysis 1: Comparison: Abdominal Aortic Aneurysm Endovascular Repair; The primary safety endpoint was tested against a predetermined safety Performance Goal (PG) using the following statistical hypotheses: H0: p ≥ 20% vs. H1: p < 20% where p is the proportion of subjects experiencing a Major Adverse Event (MAE) within 30 days of the index procedure in the target population of subjects treated with the Endurant Evo Abdominal Aortic Aneurysm (AAA) Stent graft system and 20% is the safety PG; Test type: Other; p < 0.001, Exact binomial test; Percentage = 2.9, 97.5% CI 1-sided [upper limit 8.7]

2. Primary Outcome: Primary Effectiveness Endpoint Assessed by the Number of Subjects With Technical Success at the Index Procedure.
Description: Technical success at the index procedure (as assessed intra-operatively up until closure of the access site), defined as successful delivery and deployment of the Endurant Evo AAA Stent graft system in the planned location and with no unintentional coverage of both internal iliac arteries or any visceral aortic branches and with successful removal of the delivery system
Time Frame: Index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal Aortic Aneurysm Endovascular Repair
Number analyzed (Participants) | 69
Participants | 69
Statistical Analysis 1: Comparison: Abdominal Aortic Aneurysm Endovascular Repair; The primary effectiveness endpoint was tested against a predetermined effectiveness PG using following statistical hypotheses: H0: q ≤ 80% vs. H1: q > 80% where q is the proportion of subjects who have a successful aneurysm treatment in the target population of subjects treated with the Endurant Evo AAA Stent graft system and 80% is the effectiveness PG; Test type: Other — Single-arm study with a hypothesis test comparing to performance goal; p = 0.001, Based on exact binomial distribution; Percentage = 100, 95% CI 1-sided [lower limit 95.8]

3. Secondary Outcome: Number of Subjects With All-Cause Mortality (ACM) at Each Follow up
Description: All-cause-mortality within 30, 183, and 365 days and annually until 5 years.
Time Frame: Within 30, 183, and 365 days, then annually until 5-Year post-implantation
Population: Within 0-365 days, 69 subjects were evaluable. Within 366-731 days, 66 subject were evaluable. Within 732-1096 days, 58 subjects were evaluable. Within 1097-1461 days, 50 subjects were evaluable. Within 1462-1826 days, 46 subjects were evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal Aortic Aneurysm Endovascular Repair
Number analyzed (Participants) | 69
Participants
  All-cause-mortality (ACM) 0-30 Days | 0
  All-cause-mortality (ACM) 0-183 Days | 2
  All-cause-mortality (ACM) 0-365 Days | 3
  All-cause-mortality (ACM) 366-731 Days: number analyzed (Participants) | 66
  All-cause-mortality (ACM) 366-731 Days | 3
  All-cause-mortality (ACM) 732-1096 Days: number analyzed (Participants) | 58
  All-cause-mortality (ACM) 732-1096 Days | 6
  All-cause-mortality (ACM) 1097-1461 Days: number analyzed (Participants) | 50
  All-cause-mortality (ACM) 1097-1461 Days | 1
  All-cause-mortality (ACM) 1462-1826: number analyzed (Participants) | 46
  All-cause-mortality (ACM) 1462-1826 | 3

4. Secondary Outcome: Number of Subjects With Aneurysm-related Mortality (ARM) at Each Follow up Time Point
Description: Aneurysm-related mortality within 30, 183, and 365 days, then annually until 5-Year post-implantation
Time Frame: within 30, 183, and 365 days, then annually until 5-Year post-implantation
Population: Within 0-30 days, 69 subjects were evaluable. Within 0-183 days, 69 subjects were evaluable. Within 0-365 days, 66 subjects were evaluable. Within 366-731 days, 66 subjects were evaluable. Within 732-1096 days, 58 subjects were evaluable. Within 1097-1461 days, 50 subjects were evaluable. Within 1462-1826 days, 46 subjects were evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal Aortic Aneurysm Endovascular Repair
Number analyzed (Participants) | 69
Participants
  Aneurysm-related mortality (ARM) 0-30 days | 0
  Aneurysm-related mortality (ARM) 0-183 days | 0
  Aneurysm-related mortality (ARM) 0-365 days: number analyzed (Participants) | 66
  Aneurysm-related mortality (ARM) 0-365 days | 0
  Aneurysm-related mortality (ARM) 366-731 days: number analyzed (Participants) | 66
  Aneurysm-related mortality (ARM) 366-731 days | 0
  Aneurysm-related mortality (ARM) 732-1096 days: number analyzed (Participants) | 58
  Aneurysm-related mortality (ARM) 732-1096 days | 0
  Aneurysm-related mortality (ARM) 1097-1461 days: number analyzed (Participants) | 50
  Aneurysm-related mortality (ARM) 1097-1461 days | 0
  Aneurysm-related mortality (ARM) 1462-1826 days: number analyzed (Participants) | 46
  Aneurysm-related mortality (ARM) 1462-1826 days | 0

5. Secondary Outcome: Number of Subjects With Secondary Procedures to Correct Type I and III Endoleaks Within Each Follow up Time Point
Description: Secondary procedures to correct Type I and III endoleaks within 183 and 365 day, then annually until 5-Year post-implantation
Time Frame: Within 30, 183, and 365 days, then annually until 5-Year post-implantation
Population: Within 0-30 days, 69 subjects were evaluable. Within 0-183 days, 69 subjects were evaluable. Within 0-365 days, 66 subjects were evaluable. Within 366-731 days, 65 subjects were evaluable. Within 732-1096 days, 57 subjects were evaluable. Note: Reporting of secondary endovascular procedures between 3 and 5 years of follow-up were only required when corresponding to adverse events related to the device, procedure, aneurysm, or subject death.
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal Aortic Aneurysm Endovascular Repair
Number analyzed (Participants) | 69
Participants
  0-30 Days | 0
  0-183 Days | 0
  0-365 Days: number analyzed (Participants) | 66
  0-365 Days | 1
  366-731 Days: number analyzed (Participants) | 65
  366-731 Days | 0
  732-1096 Days: number analyzed (Participants) | 57
  732-1096 Days | 1
  1097-1461 Days: number analyzed (Participants) | 51
  1097-1461 Days | 3
  1462-1826 Days: number analyzed (Participants) | 48
  1462-1826 Days | 1

6. Secondary Outcome: Number of Subjects With Secondary Endovascular Procedures Within Each Follow up Time Point
Description: Secondary endovascular procedures within 30, 183, and 365 days, then annually until 5-Year post-implantation.
Time Frame: within 30, 183, and 365 days, then annually until 5-Year post-implantation
Population: Within 0-30 days, 69 subjects were evaluable. Within 0-183 days, 69 subjects were evaluable. Within 0-365 days, 67 subjects were evaluable. Within 366-731 days, 65 subjects were evaluable. Within 732-1096 days, 57 subjects were evaluable. Within 1097-1461 Days, 50 subjects were evaluable.* Within 1462-1826 days, 46 subjects were evaluable.*
  *Reporting of events between 3 -5 years follow-up were only required when related to the device, procedure, aneurysm, or subject death
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal Aortic Aneurysm Endovascular Repair
Number analyzed (Participants) | 69
Participants
  Secondary Endovascular procedure 0-30 days | 0
  Secondary Endovascular procedure 0-183 days | 0
  Secondary Endovascular procedure 0-365 days: number analyzed (Participants) | 67
  Secondary Endovascular procedure 0-365 days | 2
  Secondary Endovascular procedure 366-731 days: number analyzed (Participants) | 65
  Secondary Endovascular procedure 366-731 days | 0
  Secondary Endovascular procedure 732-1096 days: number analyzed (Participants) | 57
  Secondary Endovascular procedure 732-1096 days | 4
  Secondary Endovascular procedure 1097- 1461 days: number analyzed (Participants) | 50
  Secondary Endovascular procedure 1097- 1461 days | 7
  Secondary Endovascular procedure 1462-1826 days: number analyzed (Participants) | 46
  Secondary Endovascular procedure 1462-1826 days | 3

7. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAE)
Description: Serious adverse events within 30, 183, and 365 days, then annually until 5-Year post-implantation
Time Frame: within 30, 183, and 365 days, then annually until 5-Year post-implantation
Population: Within 0-30 days, 69 subjects were evaluable. Within 0-183 days, 69 subjects were evaluable. Within 0-365 days, 69 subjects were evaluable. Within 366-731 days, 66 subjects were evaluable. Within 732-1096 days, 58 subjects were evaluable. Within 1097-1461 Days, 50 subjects were evaluable.* Within 1462-1826 days, 46 subjects were evaluable.*
  *Reporting of events between 3 -5 years follow-up were only required when related to the device, procedure, aneurysm, or subject death
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal Aortic Aneurysm Endovascular Repair
Number analyzed (Participants) | 69
Participants
  Serious Adverse Events (SAE) 0-30 Days | 9
  Serious Adverse Events (SAE) 0-183 Days | 19
  Serious Adverse Events (SAE) 0-365 Days | 25
  Serious Adverse Events (SAE) 366-731 Days: number analyzed (Participants) | 66
  Serious Adverse Events (SAE) 366-731 Days | 18
  Serious Adverse Events (SAE) 732- 1096 Days: number analyzed (Participants) | 58
  Serious Adverse Events (SAE) 732- 1096 Days | 19
  Serious Adverse Events (SAE) 1097-1461 Days: number analyzed (Participants) | 50
  Serious Adverse Events (SAE) 1097-1461 Days | 12
  Serious Adverse Events (SAE) 1462-1826 Days: number analyzed (Participants) | 46
  Serious Adverse Events (SAE) 1462-1826 Days | 8

8. Secondary Outcome: The Number of Subjects With Aneurysm Rupture
Description: Aneurysm rupture within 30, 183, and 365 days, then annually until 5-Year post-implantation
Time Frame: Within 30, 183, and 365 days, then annually until 5-Year post-implantation
Population: Within 0-30 days, 69 subjects were evaluable. Within 0-183 days, 69 subjects were evaluable. Within 0-365 days, 66 subjects were evaluable. Within 366-731 days, 66 subjects were evaluable. Within 732-1096 days, 58 subjects were evaluable. Within 1097-1461 Days, 49 subjects were evaluable. Within 1462-1826 days, 45 subjects were evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal Aortic Aneurysm Endovascular Repair
Number analyzed (Participants) | 69
Participants
  Aneurysm Rupture 0-30 days | 0
  Aneurysm Rupture 0-183 days | 0
  Aneurysm Rupture 0-365 days: number analyzed (Participants) | 66
  Aneurysm Rupture 0-365 days | 0
  Aneurysm Rupture 366-731 days: number analyzed (Participants) | 66
  Aneurysm Rupture 366-731 days | 0
  Aneurysm Rupture 0732-1096 days: number analyzed (Participants) | 58
  Aneurysm Rupture 0732-1096 days | 1
  Aneurysm Rupture 1097-1461 days: number analyzed (Participants) | 49
  Aneurysm Rupture 1097-1461 days | 1
  Aneurysm Rupture 1462-1826 days: number analyzed (Participants) | 45
  Aneurysm Rupture 1462-1826 days | 0

9. Secondary Outcome: The Number of Subjects With Conversion to Ppen Surgery
Description: Conversion to open surgery within 30, 183, and 365 days, then annually until 5-Year post-implantation
Time Frame: Within 30, 183, and 365 days, then annually until 5-Year post-implantation
Population: Within 0-30 days, 69 subjects were evaluable. Within 0-183 days, 69 subjects were evaluable. Within 0-365 days, 66 subjects were evaluable. Within 366-731 days, 66 subjects were evaluable. Within 732-1096 days, 58 subjects were evaluable. Within 1097-1461 Days, 50 subjects were evaluable. Within 1462-1826 days, 45 subjects were evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal Aortic Aneurysm Endovascular Repair
Number analyzed (Participants) | 69
Participants
  Conversion to open surgery 0-30 days | 0
  Conversion to open surgery 0-183 days | 0
  Conversion to open surgery 0-365 days: number analyzed (Participants) | 66
  Conversion to open surgery 0-365 days | 0
  Conversion to open surgery 365-731 days: number analyzed (Participants) | 66
  Conversion to open surgery 365-731 days | 3
  Conversion to open surgery 732-1096 days: number analyzed (Participants) | 58
  Conversion to open surgery 732-1096 days | 0
  Conversion to open surgery 1097-1461 days: number analyzed (Participants) | 50
  Conversion to open surgery 1097-1461 days | 2
  Conversion to open surgery 1462-1826 days: number analyzed (Participants) | 45
  Conversion to open surgery 1462-1826 days | 0

10. Secondary Outcome: The Number of Subjects With Major Adverse Events (MAE)
Description: Major adverse events within 183, and 365 days, then annually until 5-Year post-implantation
Time Frame: Within 183, and 365 days, then annually until 5-Year post-implantation
Population: Within 0-183 days, 69 subjects were evaluable. Within 0-365 days, 69 subjects were evaluable. Within 366-731 days, 66 subjects were evaluable. Within 732-1096 days, 58 subjects were evaluable. Within 1097-1461 Days, 50 subjects were evaluable. Within 1462-1826 days, 45 subjects were evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal Aortic Aneurysm Endovascular Repair
Number analyzed (Participants) | 69
Participants
  Major Adverse Events (MAEs) 0-183 days | 5
  Major Adverse Events (MAEs) 0-365 days | 6
  Major Adverse Events (MAEs) 366-731 days: number analyzed (Participants) | 66
  Major Adverse Events (MAEs) 366-731 days | 6
  Major Adverse Events (MAEs) 732-1096 days: number analyzed (Participants) | 58
  Major Adverse Events (MAEs) 732-1096 days | 6
  Major Adverse Events (MAEs) 1097-1461 days: number analyzed (Participants) | 50
  Major Adverse Events (MAEs) 1097-1461 days | 7
  Major Adverse Events (MAEs) 1462-1826 days: number analyzed (Participants) | 45
  Major Adverse Events (MAEs) 1462-1826 days | 5

11. Secondary Outcome: the Number of Subjects With Stent Graft Migration (as Compared to 1-month Imaging)
Description: Stent graft migration (as compared to 1-month imaging) through 12-month, 24-month, 36-month, 48-month and 60-month using worst case.
Time Frame: Through 12-month, 24-month, 36-month, 48-month and 60-month
Population: Through 12 Months, 61 subjects were evaluable. Through 24 Months, 56 subjects were evaluable. Through 36 Months, 45 subjects were evaluable. Through 48 Months, 37 subjects were evaluable. Through 60 Months, 31 subjects were evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal Aortic Aneurysm Endovascular Repair
Number analyzed (Participants) | 69
Participants
  Stent Graft Migration through 12 Months: number analyzed (Participants) | 61
  Stent Graft Migration through 12 Months | 1
  Stent Graft Migration through 24 Months: number analyzed (Participants) | 56
  Stent Graft Migration through 24 Months | 1
  Stent Graft Migration through 36 Months: number analyzed (Participants) | 45
  Stent Graft Migration through 36 Months | 1
  Stent Graft Migration through 48 Months: number analyzed (Participants) | 37
  Stent Graft Migration through 48 Months | 1
  Stent Graft Migration through 60 Months: number analyzed (Participants) | 31
  Stent Graft Migration through 60 Months | 4

12. Secondary Outcome: Number of Subjects With Aneurysm Expansion > 5 mm (as Compared to 1-month Imaging)
Description: Aneurysm expansion > 5 mm (as compared to 1-month imaging) at 12-month, 24-month, 36-month, 48-month and 60-month
Time Frame: 12-month, 24-month, 36-month, 48-month and 60-month
Population: At 12 Months, 62 subjects were evaluable. At 24 Months, 57 subjects were evaluable. At 36 Months, 43 subjects were evaluable. At 48 Months, 37 subjects were evaluable. At 60 Months, 31 subjects were evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal Aortic Aneurysm Endovascular Repair
Number analyzed (Participants) | 69
Participants
  Aneurysm Expansion at 12 Months: number analyzed (Participants) | 62
  Aneurysm Expansion at 12 Months | 1
  Aneurysm Expansion at 24 Months: number analyzed (Participants) | 57
  Aneurysm Expansion at 24 Months | 4
  Aneurysm Expansion at 36 Months: number analyzed (Participants) | 43
  Aneurysm Expansion at 36 Months | 6
  Aneurysm Expansion at 48 Months: number analyzed (Participants) | 37
  Aneurysm Expansion at 48 Months | 5
  Aneurysm Expansion at 60 Months: number analyzed (Participants) | 31
  Aneurysm Expansion at 60 Months | 2

13. Secondary Outcome: Number of Subject With Endoleaks Based on Imaging Findings
Description: Table will show a total number of subjects with endoleak at each follow up time point
Time Frame: 1- month, 6-month, 12-month, 24-month, 36-month, 48-month and 60-month
Population: At 1 Month, 66 subjects were evaluable. At 6 Months, 60 subjects were evaluable. At 12 Months, 58 subjects were evaluable. At 24 Months, 54 subjects were evaluable. At 36 Months, 40 subjects were evaluable. At 48 Months, 35 subjects were evaluable. At 60 Months, 30 subjects were evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal Aortic Aneurysm Endovascular Repair
Number analyzed (Participants) | 69
Participants
  Participants with any type of endoleak at 1 Month: number analyzed (Participants) | 66
  Participants with any type of endoleak at 1 Month | 25
  Participants with any type of endoleak at 6 Months: number analyzed (Participants) | 60
  Participants with any type of endoleak at 6 Months | 16
  Participants with any type of endoleak at 12 Months: number analyzed (Participants) | 58
  Participants with any type of endoleak at 12 Months | 14
  Participants with any type of endoleak at 24 Months: number analyzed (Participants) | 54
  Participants with any type of endoleak at 24 Months | 9
  Participants with any type of endoleak at 36 Months: number analyzed (Participants) | 40
  Participants with any type of endoleak at 36 Months | 8
  Participants with any type of endoleak at 48 Months: number analyzed (Participants) | 35
  Participants with any type of endoleak at 48 Months | 6
  Participants with any type of endoleak at 60 Months: number analyzed (Participants) | 30
  Participants with any type of endoleak at 60 Months | 2

14. Secondary Outcome: Number of Subjects With Stent Graft Occlusion Based on Imaging Findings
Description: Stent graft occlusion based on imaging findings through 6-month, 12-month, 24-month, 36-month, 48-month and 60-month
Time Frame: Through 6-month, 12-month, 24-month, 36-month, 48-month and 60-month
Population: Through 6 Months, 61 subjects were evaluable. Through 12 Months, 60 subjects were evaluable. Through 24 Months, 55 subjects were evaluable. Through 36 Months, 40 subjects were evaluable. Through 48 Months, 34 subjects were evaluable. Through 60 Months, 30 subjects were evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal Aortic Aneurysm Endovascular Repair
Number analyzed (Participants) | 69
Participants
  Stent Graft Occlusion through 6 months: number analyzed (Participants) | 61
  Stent Graft Occlusion through 6 months | 0
  Stent Graft Occlusion through 12 months: number analyzed (Participants) | 60
  Stent Graft Occlusion through 12 months | 0
  Stent Graft Occlusion through 24 months: number analyzed (Participants) | 55
  Stent Graft Occlusion through 24 months | 0
  Stent Graft Occlusion through 36 months: number analyzed (Participants) | 40
  Stent Graft Occlusion through 36 months | 0
  Stent Graft Occlusion through 48 months: number analyzed (Participants) | 34
  Stent Graft Occlusion through 48 months | 0
  Stent Graft Occlusion through 60 months: number analyzed (Participants) | 30
  Stent Graft Occlusion through 60 months | 0

15. Secondary Outcome: Number of Subject With Device Deficiencies Based on Imaging Findings
Description: Total number of subject with Any Device Deficiency through the follow up time points.
Time Frame: Through 6-month, 12-month, 24-month, 36-month, 48-month and 60-month
Population: Through 6 Months, 61 subjects were evaluable. Through 12 Months, 65 subjects were evaluable. Through 24 Months, 61 subjects were evaluable. Through 36 Months, 57 subjects were evaluable. Through 48 Months, 55 subjects were evaluable. Through 60 Months, 51 subjects were evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal Aortic Aneurysm Endovascular Repair
Number analyzed (Participants) | 69
Participants
  Any device deficiency through 6 months: number analyzed (Participants) | 61
  Any device deficiency through 6 months | 15
  Any device deficiency through 12 months: number analyzed (Participants) | 65
  Any device deficiency through 12 months | 25
  Any device deficiency through 24 months: number analyzed (Participants) | 61
  Any device deficiency through 24 months | 33
  Any device deficiency through 36 months: number analyzed (Participants) | 57
  Any device deficiency through 36 months | 35
  Any device deficiency through 48 months: number analyzed (Participants) | 55
  Any device deficiency through 48 months | 36
  Any device deficiency through 60 months: number analyzed (Participants) | 51
  Any device deficiency through 60 months | 36

ADVERSE EVENTS:
Time Frame: 60-months
Arm/Group | Abdominal Aortic Aneurysm Endovascular Repair
All-Cause Mortality (participants affected / at risk) | 16/69
Serious Adverse Events (participants affected / at risk) | 54/69
Other Adverse Events (participants affected / at risk) | 6/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abdominal Aortic Aneurysm Endovascular Repair (N=69)
ANGINA PECTORIS (Cardiac disorders) | 2 (2)
ANGINA UNSTABLE (Cardiac disorders) | 2 (3)
AORTIC VALVE STENOSIS (Cardiac disorders) | 1 (1)
BRADYCARDIA (Cardiac disorders) | 2 (2)
CARDIAC ARREST (Cardiac disorders) | 3 (3)
CARDIAC FAILURE (Cardiac disorders) | 1 (1)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 (1)
SICK SINUS SYNDROME (Cardiac disorders) | 1 (1)
HYDROCELE (Congenital, familial and genetic disorders) | 1 (1)
CATARACT (Eye disorders) | 1 (1)
DIVERTICULUM (Gastrointestinal disorders) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1)
INTESTINAL POLYP (Gastrointestinal disorders) | 1 (1)
LOCALISED INTRAABDOMINAL FLUID COLLECTION (Gastrointestinal disorders) | 1 (1)
SMALL INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
ASTHENIA (General disorders) | 1 (1)
DEATH (General disorders) | 2 (2)
DEVICE DAMAGE (General disorders) | 1 (1)
DEVICE DISLOCATION (General disorders) | 1 (1)
PYREXIA (General disorders) | 1 (1)
STENT-GRAFT ENDOLEAK (General disorders) | 8 (9)
THROMBOSIS IN DEVICE (General disorders) | 2 (4)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 2 (2)
BACTERIAL INFECTION (Infections and infestations) | 2 (2)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (1)
GROIN INFECTION (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 3 (3)
PNEUMONIA LEGIONELLA (Infections and infestations) | 1 (1)
POSTOPERATIVE ABSCESS (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
UROSEPSIS (Infections and infestations) | 1 (1)
CARBON MONOXIDE POISONING (Injury, poisoning and procedural complications) | 1 (1)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
CONCUSSION (Injury, poisoning and procedural complications) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1 (2)
PERIPHERAL ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 1 (1)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1)
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1)
BLOOD POTASSIUM DECREASED (Investigations) | 1 (1)
PROPOFOL INFUSION SYNDROME (Metabolism and nutrition disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 1 (1)
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 1 (1)
ACUTE LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
MALIGNANT NEOPLASM OF RENAL PELVIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
METASTATIC SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
NASAL NEOPLASM BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
NON-HODGKIN'S LYMPHOMA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
NON-SMALL CELL LUNG CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PROSTATE CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
RECURRENT CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
CAROTID ARTERIOSCLEROSIS (Nervous system disorders) | 1 (1)
CEREBRAL INFARCTION (Nervous system disorders) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1)
NEUROLOGICAL SYMPTOM (Nervous system disorders) | 1 (1)
NEUROTOXICITY (Nervous system disorders) | 1 (1)
PARKINSON'S DISEASE (Nervous system disorders) | 2 (2)
PETIT MAL EPILEPSY (Nervous system disorders) | 1 (1)
ANXIETY (Psychiatric disorders) | 2 (2)
DEPRESSION (Psychiatric disorders) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 1 (1)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 2 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (2)
PHARYNGEAL HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 (2)
HIP ARTHROPLASTY (Surgical and medical procedures) | 1 (1)
ANEURYSM (Vascular disorders) | 2 (2)
AORTIC ANEURYSM RUPTURE (Vascular disorders) | 2 (2)
HAEMORRHAGE (Vascular disorders) | 1 (1)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 (1)
PERIPHERAL ARTERY STENOSIS (Vascular disorders) | 1 (1)
PERIPHERAL ARTERY THROMBOSIS (Vascular disorders) | 2 (2)
THROMBOSIS (Vascular disorders) | 2 (2)
VASCULAR STENOSIS (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abdominal Aortic Aneurysm Endovascular Repair (N=69)
PYREXIA (General disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-07-26): https://cdn.clinicaltrials.gov/large-docs/24/NCT02461524/Prot_000.pdf
  • Statistical Analysis Plan (2015-05-04): https://cdn.clinicaltrials.gov/large-docs/24/NCT02461524/SAP_001.pdf